CLINICAL TRIAL: NCT03906916
Title: Multicenter Study to Compare Two Diagnostic Tests (1,3-β-D-glucan vs Blood Culture) in Critically Ill Patients With Suspected Invasive CAndidiasis Hospitalized in Internal Medicine Wards and Who Are Currently Timely Treated With Echinocandin (Micafungin)
Brief Title: Comparison of Two Diagnostic Tests in Patients With Suspected Invasive Candidiasis in Internal Medicine Wards and Who Are Currently Timely Treated With Micafungin
Acronym: EPICA1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was interrupted prematurely because of the low rate of recruitment.
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FADOI.02.2017
Record Dates: First submitted 2018-07-20; First posted 2019-04-08 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Invasive Candidiasis
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspicion of invasive candidiasis (Experimental): Patients hospitalised in Internal Medicine with suspicion of invasive candidiasis will be treated with an echinocandin (micafungin) as timely as possible, and they will continue the antifungal treatment according to international guidelines when diagnosis is confirmed by positive 1,3-β-D-glucan test.
  Interventions: Diagnostic Test: 1,3-β-D-glucan quantification; Drug: Micafungin

INTERVENTIONS:
Diagnostic Test: 1,3-β-D-glucan quantification — Patients hospitalised in Internal Medicine with suspicion of invasive candidiasis will be evaluated by 1,3-β-D-glucan test and by means of blood culture to confirm the diagnosis
  Other Names: FUNGITELL
Drug: Micafungin — Patients hospitalised in Internal Medicine with suspicion of invasive candidiasis will be treated with an echinocandin (micafungin) as timely as possible, and they will continue the antifungal treatment according to international guidelines when diagnosis is confirmed by positive 1,3-β-D-glucan test.

SUMMARY:
EPICA-1 is a multicenter, open label, interventional study which will involve about 30 Internal Medicine Units throughout Italy, enrolling globally at least 100 hospitalised patients with suspicion of invasive candidiasis. These patients will be treated with an echinocandin (micafungin) as timely as possible, and they will continue the antifungal treatment according to international guidelines when diagnosis is confirmed by positive 1,3-β-D-glucan test: this will allow collection of information on patients outcome. At the same time, patients will be also evaluated by means of blood culture, so that comparison will be possible between the two diagnostic tests (primary end-point of the study).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Patients giving their informed consent to participate to the study and to the use of their health data
* Patients with two or more SIRS criteria (hyperthermia, or hypothermia, tachycardia, tachypnea, leucocytosis or leukopenia )
* Patients treated with antibiotic therapy in the last 4 weeks and with central venous catheter
* Patients with at least one of these conditions ( cortisone therapy/ immunosuppressive agents, total parenteral nutrition, urinary catheter, anticancer chemotherapy and major surgery in the last 3 weeks, acute pancreatitis, diabetes mellitus, liver diseases, dialysis)

Exclusion Criteria:

* Patients with ALT, AST, bilirubin > 3 times the upper limit of normal
* Patients enrolled in other interventional clinical studies
* Patients treated with echinocandin or azolic or polyene at the time of the enrolment
* Pregnancy or breastfeeding
* Neutropenic patients
* HIV positive patients
* Central nervous system events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
To assess the equivalence between two diagnostic test for Candida infections: 1,3-β-D-glucan vs. emocoltura | 14 days
  Will be compared the results of the two diagnostic tests for the same patient's blood sample. In particular will be evaluated if there is accordance between the Candida positivity of an emocolture and the positivity of the 1,3-β-D-glucan test (1,3-β-D-glucan concentrations > 200 pg/ml) for the same patient's blood sample.

SECONDARY OUTCOMES:
To assess the effect of a pre-emptive micafungin treatment on the outcome of patients. | 14 days
  Will be evaluated the mortality (number of dead patients) and ICU transfering (number of patients move to the ICU) reductions
To describe the trend of 1,3-β-D-glucan in patients during micafungin treatment | 14 days
  Will be measured the 1,3-β-D-glucan concentrations in in patients during micafungin treatment

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - Osp. Generale Regionale F. Miulli, Acquaviva delle Fonti
  - Nuovo Ospedale Civile S. Agostino-Estense, Baggiovara
  - Ospedale di Bussolengo, Bussolengo
  - Ospedale "S. Anna", Castelnovo ne' Monti
  - ASL CN1 Ospedale di Ceva, Ceva
  - Ospedale Maggiore, Chieri
  - Ospedale "S. Anna", Como
  - Ospedale "S. Biagio", Domodossola
  - Ente Ospedaliero Galliera, Genova
  - Ospedale "Mater Salutis", Legnago
  - Ospedale "S.M. Bianca", Mirandola
  - Ospedale di Mondovì,, Mondovì
  - Ospedale "Antonio Cardarelli, Napoli
  - Presidio Ospedaliero S. Maria Delle Grazie, Pozzuoli
  - Ospedale "G. Fracastoro", San Bonifacio
  - Nuovo Ospedale Civile di Sassuolo, Sassuolo
  - Ospedale Maggiore SS. Annunziata, Savigliano
  - Ospedale Civile di Sestri Levante, Sestri Levante
  - Policlinico Borgo Roma, Verona
  - Ospedale "Magalini, Villafranca di Verona